CLINICAL TRIAL: NCT03350945
Title: Application of Carbon Nanoparticles in Laparoscopic Colorectal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aiguo, Lu (Other)
Responsible Party: Sponsor-Investigator, Aiguo, Lu, Clinical Professor, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LAiguo
Record Dates: First submitted 2017-11-05; First posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Colorectal Tumor
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Device:Titanium Clips (Active Comparator): Device: Tumor localization. Preoperative endoscopic localization with titanium clips
  Interventions: Procedure: Device: tumor localization
- Device:Intra-operative Endoscopy (Active Comparator): Device: Tumor localization. During the laparoscopic surgery,tumor is localized using intra-operative endoscopy detection.
  Interventions: Procedure: Device: tumor localization
- Device:Carbon Nanoparticles (Experimental): Device: Tumor localization. During the laparoscopic surgery,tumor is localized using carbon nanoparticles.
  Interventions: Procedure: Device: tumor localization

INTERVENTIONS:
Procedure: Device: tumor localization — At present, three dominant methods can be available to locate tumor: preoperative endoscopic clip placement, intraoperative endoscopy and endoscopic tattooing

SUMMARY:
The project aims to evaluate the safety, effectiveness, accuracy and economy efficiency of the application of carbon nanoparticles for tumor localization and lymph nodes mapping in the laparoscopic coloectal surgery.

DETAILED DESCRIPTION:
Colorectal cancer is among the most commonly diagnosed cancer in both men and women . Increasing studies have been focused on the causes and therapies of this disease in order to improve the prognosis. In recent decades, laparoscopy has been commonly used in both colorectal and gastric surgery due to the benefit of minimal invasive technology progression . Its comparable safety and effectiveness have been proved in many studies. The advantages of minimal invasive surgery such as faster recovery, less bleeding and less pain, have also been admitted by numerous surgeons . However, the accomplishment of operation procedures mainly depend on subjective experiences. Even skilled surgeons can be impeded in operation due to the deficiency of tactile sense . As a result, accurate intra-operative localization of tumor would be a tough task if it was invisible on the serosal surface or difficult to approach, such as small or flat neoplasms, tumor confined to the mucosa and submucosa and endoscopically resected polyps which required additional surgery . At present, three dominant methods can be available to locate tumor: preoperative endoscopic clip placement, intraoperative endoscopy and endoscopic tattooing. All of these methods have their advantages but also some unavoidable limitations, such as localization error and problems in the assessment of incision margin using preoperative clip placement, unsatisfactory operation exposure after intraoperative endoscopy, ink spillage or failure in finding lesions with dye endoscopic injection et al. Usually surgeons choose different methods according to the objective conditions such as the ability to perform endoscopy or the availability of suitable tattooing material.

Apart from the precise localization of tumor, adequate lymph node dissection is another crucial point in colorectal operation. According to AJCC recommendation and NCCN guideline, the number of lymph nodes, which has been proved of prognostic and therapeutic importance, is clearly defined in colorectal cancer to make sure of the accurate pathological staging. Previous studies have found that the number of lymph nodes evaluated after surgical resection was positively associated with the survival of patients. Besides Total Mesorectal Excision (TME) and D3 lymph node clearance, which are standards in colorectal surgery over decades of research and accumulated data, the harvest of lymph nodes is still associated with pathological doctors' experience and pathological examination skills. However, population-based data suggest that lymph node evaluation is not adequate in the majority of patients . Some micro lymph nodes, especially with diameter less than 5 mm, are more easily missed in specimen process while rate of metastasis is comparably higher in these lymph nodes. As a result, clinicians are trying to find a lymph node tracer to help improve the amount of lymph node harvest as well as the rate of micro-metastasis in lymph node.

Carbon nanoparticle has been used as a lymph node tracer for decades. As a lymphatic vessel specific dye material, there is no doubt in its effect on lymph node mapping. In recent years, surgeons have applied this tracer widely in breast and thyroid operations for sentinel lymph node mapping to determine dissection extent. The effectiveness and accuracy of this method has been verified in thyroid and breast surgery while there is rare study focused on its application in colorectal surgery. The application of tattooing material, such as methylene blue, India ink and nano-materials in tumor localization has also attracted attentions of clinicians. In our study, three groups based on different tumor localization means are compared on short-term benefits, cost-effectiveness and lymph node clearance in order to choose the best approach to locate tumor and validate lymph node staining effect of carbon nanoparticles.

ELIGIBILITY:
Inclusion Criteria:

- Pathologically diagnosed as colorectal benign tumor or tumor with TNM staging I-III (including patients need further surgery after endoscopic treatment), Be able to tolerate laparoscopic radical resection With normal hepatic and renal function No history of abdominal surgery

Exclusion Criteria:

- Patients with distant metastasis, poor compliance, prior abdominal surgery Emergency case with obstruction or perforation Have received neoadjuvant chemotherapy or radiotherapy Patients diagnosed as familial adenomatous polyposis (FAP), Inflammatory bowel disease such as ulcerative colitis and Crohn's disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor localization time | within 1 month
  From abdominal exploration to tumor localization

SECONDARY OUTCOMES:
survival data 1 | within 5 year
  overall survival
survival data 2 | within 5 year
  disease free survival
Post-operative complication rates | within 6 month
  According to the records in hospital
Distal edge distance of specimen | within 2 weeks
  measured by two pathologists separately
LN number dissected | within 2-3 weeks
  measured by two pathologists separately
Length of stay | within a year
  According to the record in hospital
Total operation time | within 1 week
  Measured according to operation record
Blood loss | within 1 week
  Measured according to operation record

CONTACTS AND LOCATIONS:
Overall Officials: Minhua Zheng, Study Chair — Ruijin Hospital

IPD SHARING:
Plan to Share IPD: Undecided